CLINICAL TRIAL: NCT04283604
Title: The Effects of a Single Dose of Methylphenidate on Motor Performance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loewenstein Hospital (Other)
Collaborators: Tel Aviv University (Other); Wingate Institute (Other)
Responsible Party: Principal Investigator, Aviva Mimouni-Bloch, Head of child developmental center, Loewenstein Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 0007-19-LOE
Record Dates: First submitted 2020-02-22; First posted 2020-02-25 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: ADHD
Keywords: Concerta; Physical Activity; Motor test; Exercise; Ritalin
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity | interventions — 5,10-dihydro-5-methylphenazine; Methylphenidate

STUDY DESIGN:
Intervention Model Description: The study will be divided into two sub studies (100 participants each), in which 50 ADHD and 50 non-ADHD participants will be included. In the first session, all participants will undergo motor tests, in the same conditions. In the second session, half of ADHD participants (25) will be asked to take their regular MPH treatment, before the session. All other participants (25 ADHD and 50 non-ADHD) will perform the motor tests without treatment, and serve as control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ADHD with MPH (Experimental): ADHD participants, taking MPH before the second session
  Interventions: Drug: MPH
- ADHD no MPH (No Intervention): ADHD participants will perform motor tests in both session, without any intervention, for evaluation of learning effect among ADHD participants.
- Healthy participants (No Intervention): Non-ADHD participants will serve as a control group for learning effect on motor tests

INTERVENTIONS:
Drug: MPH — The treatment will include taking the patient's own medication by the patient himself in the treatment session 60-180 minutes before the beginning of the tests, according to their prescription given by their own physician. Participants must have consumed this medication at least 3 months before the first session as their regular treatment for ADHD. Note, we are not planning on giving the medication to the participant, rather he/she will consume their own prescribed MPH by them self.
  Other Names: Concerta; Ritalin
  Arms: ADHD with MPH

SUMMARY:
Aim: To evaluate the effects of MPH on young adults diagnosed with ADHD on different exercise performance tests.

Hypothesis: MPH will have positive effects on motor tests requiring concentration.

Methods: 200 healthy physical education students, 100 participants diagnosed with ADHD will serve as the treatment group and 100 non-ADHD diagnosed will serve as a control group. The study will be divided into two sub studies (100 participants each), in which, two motor tests will be evaluated (two agility tests, two motor accuracy tests and balance).

All participants will arrive for two sessions, and will perform two motor tests in each session. In the second session, half of the participants with ADHD (25 participants) will undergo another session of the same motor tests with their usual treatment (treatment group) and another half (25 participants) without their treatment (ADHD control group). The non-ADHD control group (50 participants) will perform the second session without medications - to assess a learning effect.

Note, the investigators are not planning on giving the medication to the participant, rather he/she will consume their own prescribed MPH by them self. Control treatment for ADHD participants will consist of not taking their medication before the motor test.

For evaluation of physiological responses and perception of effort, heart rate, temperature, blood pressure and RPE before and after motor tests, will be measured.

DETAILED DESCRIPTION:
200 healthy physical education students and Mechina from the Academic College at Wingate, males and females, will be recruited to the study. 100 participants diagnosed with ADHD will serve as the treatment group and 100 non-ADHD diagnosed will serve as a control group.

Recruitment procedure will consist of emails to all students in college or by entering classes or zoom meetings. Volunteers answering the mail or providing their contact details will be regarded as giving consent to be addressed by the research assistant by a phone call. A research assistant will call volunteers and will briefly explain the study procedures and invite them to the first session in which they will sign an informed consent form approved by the institutional review board (Helsinki). Next, all participants will fill a general background questionnaire and an ADHD self-report scale questionnaire.

The second and third sessions will consist of motor tests, at least one week apart. In one of the sessions, ADHD volunteers will kindly be asked to arrive to the session before they took their stimulant medication or to come to the session after consuming their usual treatment (1 hour before the session begins). The order of sessions with or without treatment will be randomly decided. The investigators point out that the patient takes his own treatment himself when assigned to the ADHD treatment group. The non-ADHD control group (50 participants) will perform the two sessions without medications - to assess a learning effect.

The background questionnaire consists of general information relevant for the study. This includes name, gender, anthropometrical characteristics, chronic illness, regular medication consumption, etc. In addition, the participant will answer questions regarding diagnosis of ADHD, MPH consumption and physical activity participation.

The participants will fill the Adult ADHD Self Report Screen (ASRS) in Hebrew. This form was shown to be valid, reliable and had good internal consistence. This screen will be used for correlation analysis oh ADHD severity and exercise performance. The form is attached in this proposal.

The treatment will include taking the patient's own medication by the patient himself in the treatment session 60-180 minutes before the beginning of the tests, according to their prescription given by their own physician. Participants must have consumed this medication at least 3 months before the first session as their regular treatment for ADHD. Note, the investigators are not planning on giving the medication to the participant, rather he/she will consume their own prescribed MPH by them self.

Control treatment for ADHD participants will consist of not taking their medication before the motor test. Since there may be participant who needs to take the medication every day, they will be instructed to consume their medication at the end of the session. In this case, session meeting will be performed at morning time.

Motor tests Balance test One-leg blind balance test will be performed. The maximum number of seconds a participant is able to stand without toppling or putting a foot down will be noted. Participants will stand on both legs with eyes open, facing forward, and then lift one leg with eyes closed, facing forward on a marked site. Time recording will be stopped when participants will begin to teeter; put the foot on the floor or open their eyes. Two attempts (one for each leg) will be made, and the higher value of these two attempts will be used.

Agility tests Two agility tests will be performed twice, the best time of each test will be recorded. Calculation of the ratio of zigzag test without the ball and with the ball will be conducted on a sports hall. These two agility tests were evaluated and validated elsewhere.

Zigzag test- Running agility test. Participant is required to run a course in the shortest possible time A zigzag course consists of a rectangle 3 X 5 meters set out at 100º angles by four cones placed on the corners, with one more cone placed in the center (Fig 1). Overall there are 6 segments numbered from 1-6 according to their order in the test. This test measures rapid acceleration, deceleration and balance control

Fig 1. Schematic representation of the Zigzag Test. Noted the start and stop points. The pathways are indicated as arrows and are numbered according to their order in the test. Triangles indicates cones.

Zigzag with a ball- The same as the former test (fig 1), but with a ball. Participants will be instructed to run as fast as possible with the ball. This test measures rapid acceleration, deceleration and balance control as well as controlling the ball.

Accuracy motor tests The stationary free throw shooting test- Each participant will perform three series of ten free-throw shots (two throws in five different positions) with a 3-minute rest period between the series. Two participants will be positioned below the hoop and they will pass the ball to the testee. After the participant completes ten shots, another participant will come to the free throw line and will perform the same task. The average scores of the all three trials will be used for analysis.

Fig 2. Schematic representation of the stationary free throw shooting test. Arrows indicate shooting positions. Order of the throwing positions are numbered.

The dynamic 60-second free throw shooting test- For easier organization of the testing a volleyball court will be used as illustrated in Figure 1. Each participant will perform five series of two free throws with sprinting between the series. Each series will be completed in 12 seconds. Each participant will start the test with an 18-meter sprint (volleyball court sideline), then will turn around a cone and run to the free throw line. After performing two free throws the participant will run to another cone where he will wait for a sound signal to start the next series. One tester will use a stopwatch to measure 12 seconds, and to give a signal to the participant. Another tester will count the number of free throws made. Two other participants will pass the balls to the testee. The participants will perform the three dynamic tests with a five-minute recovery between each. The average scores of all three trials will be used for analysis.

Fig 2. The dynamic 60-second free throw shooting test.

Measurements Blood pressure- blood pressure will be measured at the beginning of each session. Peak BP will be measured at the end of the last motor test at each session. BP will be measured by using a mercury sphygmomanometer.

Body temperature- body temperature will be measured sublingually at the beginning of each session. Peak BP will be measured at the end of the last motor test at each session. Temperature will be measured by using an electronic thermometer.

Heart rate- resting heart rates will be recorded at the beginning of each session, and at the end of the last motor test. HR will be measured by a polar watch (Polar heart rate monitor S 710).

RPE scale- To measure subjective sense of effort the Borg rate of perceived exertion (RPE) scale (ranges from 6 to 20) will be used at the end of the last motor test at each session.

ELIGIBILITY:
Inclusion Criteria:

Students age 18-45 years old studying at the academic college at Wingate. For the treatment group we will recruit students who were previously diagnosed by a neurologist or psychiatrist or other ADHD physician specialist as having ADHD, and are treated with a methylphenidate (Ritalin; Ritalin SR; Ritalin LA; Concerta) at least 3 months before the first session. Control group will consist of students without ADHD.

Exclusion Criteria:

any chronic illness other than ADHD (e.g. asthma, gastrointestinal, depression, anxiety, etc.), taking chronic medications apart from stimulant therapy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Agility tests | 2 min
  Two agility tests (Zigzag with and without a ball) will be performed. The best time of each test will be recorded. Calculation of the ratio of zigzag test without the ball and with the ball will be conducted
Accuracy motor tests | 10 min
  Two accuracy motor tests (the stationary free throw shooting test and the dynamic 60-second free throw shooting test) will be performed three times. The average scores of the all three trials will be used for analysis.

SECONDARY OUTCOMES:
Blood pressure (BP) | 1 min X 2 times
  BP will be measured before and after motor test by using a mercury sphygmomanometer.
Body Temperature | 1 min X 2 times
  body temperature will be measured sublingually at the beginning and at the end of each motor test using an electronic thermometer
Heart rate (HR) | Continuously for 10 min
  Heart rates will be continuously recorded throughout the test (Polar heart rate monitor S 710). HR before and after the tests will be recorded
Rate of Perceived exertion (RPE) scale | 10 sec X 2 times
  To measure subjective sense of effort we will use the Borg rate of perceived exertion (RPE) scale (ranges from 6 to 20) at the end of each motor test.

CONTACTS AND LOCATIONS:
Locations (1):
- Sharon Tsuk, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Battle DE. Diagnostic and Statistical Manual of Mental Disorders (DSM). Codas. 2013;25(2):191-2. doi: 10.1590/s2317-17822013000200017. No abstract available. PMID 24413388
- [Background] Huss M, Duhan P, Gandhi P, Chen CW, Spannhuth C, Kumar V. Methylphenidate dose optimization for ADHD treatment: review of safety, efficacy, and clinical necessity. Neuropsychiatr Dis Treat. 2017 Jul 4;13:1741-1751. doi: 10.2147/NDT.S130444. eCollection 2017. PMID 28740389
- [Background] Zimmer L. Contribution of Clinical Neuroimaging to the Understanding of the Pharmacology of Methylphenidate. Trends Pharmacol Sci. 2017 Jul;38(7):608-620. doi: 10.1016/j.tips.2017.04.001. Epub 2017 Apr 24. PMID 28450072
- [Background] Shorer Z, Bachner Y, Guy T, Melzer I. Effect of single dose methylphenidate on walking and postural stability under single- and dual-task conditions in older adults--a double-blind randomized control trial. J Gerontol A Biol Sci Med Sci. 2013 Oct;68(10):1271-80. doi: 10.1093/gerona/glt035. Epub 2013 Apr 11. PMID 23580740
- [Background] Ben-Itzhak R, Giladi N, Gruendlinger L, Hausdorff JM. Can methylphenidate reduce fall risk in community-living older adults? A double-blind, single-dose cross-over study. J Am Geriatr Soc. 2008 Apr;56(4):695-700. doi: 10.1111/j.1532-5415.2007.01623.x. Epub 2008 Feb 7. PMID 18266665
- [Background] Cordeiro LMS, Rabelo PCR, Moraes MM, Teixeira-Coelho F, Coimbra CC, Wanner SP, Soares DD. Physical exercise-induced fatigue: the role of serotonergic and dopaminergic systems. Braz J Med Biol Res. 2017 Oct 19;50(12):e6432. doi: 10.1590/1414-431X20176432. PMID 29069229
- [Background] King M, Rauch LHG, Brooks SJ, Stein DJ, Lutz K. Methylphenidate Enhances Grip Force and Alters Brain Connectivity. Med Sci Sports Exerc. 2017 Jul;49(7):1443-1451. doi: 10.1249/MSS.0000000000001252. PMID 28277403
- [Background] Swart J, Lamberts RP, Lambert MI, St Clair Gibson A, Lambert EV, Skowno J, Noakes TD. Exercising with reserve: evidence that the central nervous system regulates prolonged exercise performance. Br J Sports Med. 2009 Oct;43(10):782-8. doi: 10.1136/bjsm.2008.055889. Epub 2008 Dec 3. PMID 19052141
- [Background] Roelands B, Hasegawa H, Watson P, Piacentini MF, Buyse L, De Schutter G, Meeusen RR. The effects of acute dopamine reuptake inhibition on performance. Med Sci Sports Exerc. 2008 May;40(5):879-85. doi: 10.1249/MSS.0b013e3181659c4d. PMID 18408610
- [Background] Marcora S. Can Doping be a Good Thing? Using Psychoactive Drugs to Facilitate Physical Activity Behaviour. Sports Med. 2016 Jan;46(1):1-5. doi: 10.1007/s40279-015-0412-x. No abstract available. PMID 26497149
- [Background] Stray LL, Ellertsen B, Stray T. Motor function and methylphenidate effect in children with attention deficit hyperactivity disorder. Acta Paediatr. 2010 Aug;99(8):1199-204. doi: 10.1111/j.1651-2227.2010.01760.x. Epub 2010 Mar 12. PMID 20298494
- [Background] Klass M, Roelands B, Levenez M, Fontenelle V, Pattyn N, Meeusen R, Duchateau J. Effects of noradrenaline and dopamine on supraspinal fatigue in well-trained men. Med Sci Sports Exerc. 2012 Dec;44(12):2299-308. doi: 10.1249/MSS.0b013e318265f356. PMID 22776872
- [Background] Kang KD, Yun SW, Chung U, Kim TH, Park JH, Park IH, Han DH. Effects of methylphenidate on body index and physical fitness in Korean children with attention deficit hyperactivity disorder. Hum Psychopharmacol. 2016 Mar;31(2):76-82. doi: 10.1002/hup.2514. Epub 2016 Jan 12. PMID 26756111
- [Background] Bart O, Daniel L, Dan O, Bar-Haim Y. Influence of methylphenidate on motor performance and attention in children with developmental coordination disorder and attention deficit hyperactive disorder. Res Dev Disabil. 2013 Jun;34(6):1922-7. doi: 10.1016/j.ridd.2013.03.015. Epub 2013 Apr 10. PMID 23584172
- [Background] Meckel Y, Nemet D, Eliakim A. the Effect of Methylphenidate Treatment on Exercise Performance in Children With Attention-Deficit Hyperactivity Disorder. Acta Kinesiol. Univ. Tartu 7:109-16, 2011
- [Background] De Crescenzo F, Armando M, Mazzone L, Ciliberto M, Sciannamea M, Figueroa C, Janiri L, Quested D, Vicari S. The use of actigraphy in the monitoring of methylphenidate versus placebo in ADHD: a meta-analysis. Atten Defic Hyperact Disord. 2014 Mar;6(1):49-58. doi: 10.1007/s12402-013-0122-x. Epub 2013 Nov 28. PMID 24287735
- [Background] Edvinsson D, Ekselius L. Long-Term Tolerability and Safety of Pharmacological Treatment of Adult Attention-Deficit/Hyperactivity Disorder: A 6-Year Prospective Naturalistic Study. J Clin Psychopharmacol. 2018 Aug;38(4):370-375. doi: 10.1097/JCP.0000000000000917. PMID 29927781
- [Background] Zohar AH, Konfortes H. Diagnosing ADHD in Israeli adults: the psychometric properties of the adult ADHD Self Report Scale (ASRS) in Hebrew. Isr J Psychiatry Relat Sci. 2010;47(4):308-15. PMID 21270505
- [Background] Mirkov D, Nedeljkovic A, Kukolj M, Ugarkovic D, Jaric S. Evaluation of the reliability of soccer-specific field tests. J Strength Cond Res. 2008 Jul;22(4):1046-50. doi: 10.1519/JSC.0b013e31816eb4af. PMID 18545209
- [Background] Masuda S, Suganuma K, Kaneko C, Hoshina K, Suzuki T, Serita T, Sakakibara R. Prediction of Falls Using a 3-m Zigzag Walk Test. J Phys Ther Sci. 2013 Sep;25(9):1051-4. doi: 10.1589/jpts.25.1051. Epub 2013 Oct 20. PMID 24259913
- [Background] Aquino R, Palucci Vieira LH, de Paula Oliveira L, Cruz Goncalves LG, Pereira Santiago PR. Relationship between field tests and match running performance in high-level young Brazilian soccer players. J Sports Med Phys Fitness. 2018 Mar;58(3):256-262. doi: 10.23736/S0022-4707.17.06651-8. Epub 2017 Feb 14. PMID 28198600
- [Background] Archer DT, Drysdale K, Bradley EJ. Differentiating technical skill and motor abilities in selected and non-selected 3-5 year old team-sports players. Hum Mov Sci. 2016 Jun;47:81-87. doi: 10.1016/j.humov.2016.02.001. Epub 2016 Feb 22. PMID 26904973
- [Background] Pojskic H, Muratovic M. The relationship between physical fitness and shooting accuracy of professional basketball players 20:1-13, 2014
- [Background] Borg GA. Perceived exertion. Exerc Sport Sci Rev. 1974;2:131-53. No abstract available. PMID 4466663